CLINICAL TRIAL: NCT00543569
Title: A Phase 2, Randomized, Open-Label, Parallel Group, Multi-Center Study to Assess the Safety and Efficacy of Alefacept in de Novo Kidney Transplant Recipients
Brief Title: A Study to Assess the Safety and Efficacy of Alefacept in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0485-CL-U201
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Transplantation
Keywords: kidney transplant; alefacept
MeSH Terms: interventions — Alefacept; Tacrolimus; Basiliximab; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tacrolimus/MMF/Basiliximab (Active Comparator): Participants received tacrolimus at a starting dose of 0.20 mg/kg/day, mycophenolate mofetil (MMF) 750 or 1000 mg twice daily (BID), basiliximab administered as a 20 mg bolus injection 2 hours prior to transplantation on Day 0 and a 20 mg bolus injection on Day 3 and tapered corticosteroids for 6 months.
  Interventions: Drug: tacrolimus; Drug: basiliximab; Drug: mycophenolate mofetil; Drug: Corticosteroids
- Alefacept QW/Tacrolimus/MMF (Experimental): Participants received alefacept administered as a 7.5 mg intravenous (IV) bolus on Days 0 and 3; 15 mg subcutaneously on Day 7 then weekly (QW) for 12 weeks, then 15 mg subcutaneously monthly until the end of month 6, in addition to tacrolimus at a starting dose of 0.10 mg/kg/day, MMF 750 or 1000 mg BID and tapered corticosteroids for 6 months.
  Interventions: Drug: Alefacept; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: Corticosteroids
- Alefacept QW/Tacrolimus (Experimental): Participants received alefacept administered as a 7.5 mg IV bolus on Days 0 and 3; 15 mg subcutaneously on Day 7 then weekly for 12 weeks, then 15 mg subcutaneously monthly until the end of month 6, in addition to tacrolimus at a starting dose of 0.20 mg/kg/day, and tapered corticosteroids for 6 months.
  Interventions: Drug: Alefacept; Drug: tacrolimus; Drug: Corticosteroids
- Alefacept QOW/Tacrolimus/MMF (Experimental): Participants received alefacept administered as a 7.5 mg IV bolus on Days 0 and 3; 30 mg subcutaneously on Day 7 then weekly for 12 weeks, then 15 mg subcutaneously monthly until the end of month 6, in addition to tacrolimus at a starting dose of 0.10 mg/kg/day, MMF 750 or 1000 mg BID, and tapered corticosteroids for 6 months.
  Interventions: Drug: Alefacept; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: Corticosteroids

INTERVENTIONS:
Drug: Alefacept — Administered as a 7.5 mg intravenous bolus on day 0 (intraoperatively, prior to kidney revascularization) and Day 3; subsequently administered subcutaneously either weekly or every 2 weeks.
  Other Names: Amevive, ASP0485
  Arms: Alefacept QOW/Tacrolimus/MMF; Alefacept QW/Tacrolimus; Alefacept QW/Tacrolimus/MMF
Drug: tacrolimus — The initial dose of tacrolimus was administered orally within 48 hours post-transplant. Subsequent doses were to be adjusted to achieve target whole blood trough concentrations.
  Other Names: Prograf, FK506
Drug: basiliximab — Administered as a 20 mg bolus injection within 2 hours prior to transplantation and a 20 mg bolus injection on Day 3.
  Other Names: Simulect
  Arms: Tacrolimus/MMF/Basiliximab
Drug: mycophenolate mofetil — Administered at 750 mg twice per day orally or intravenously for patients enrolled under Amendment 6 or earlier and at 1000 mg twice per day orally or intravenously for patients enrolled under Amendment 7. The dose of MMF could be adjusted based on clinical symptoms.
  Other Names: CellCept, MMF
  Arms: Alefacept QOW/Tacrolimus/MMF; Alefacept QW/Tacrolimus/MMF; Tacrolimus/MMF/Basiliximab
Drug: Corticosteroids — Corticosteroids were administered as a 500 to 1000 mg intravenous bolus on Day 0 and a 125 to 250 mg methylprednisone (or equivalent oral/intravenous corticosteroid dose) on Day 1. Oral prednisone was to be tapered per protocol.

SUMMARY:
A study to assess the safety and efficacy of Alefacept in de novo kidney transplant patients.

DETAILED DESCRIPTION:
This is a 4 arm (all active) study to determine the safety and efficacy of Alefacept in de novo kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is anticipated to receive first oral dose of tacrolimus within 48 hours of transplant procedure
* Subject is a recipient of a de novo kidney transplant
* Subject is a recipient of a kidney from a non-human leukocyte antigen (HLA) identical related living donor, a non-related living donor, or a deceased donor

Exclusion Criteria:

* Subject has a screening (pre-operative)estimated cluster of differentiation (CD) 4+ T-cell count of < 250 cells/µL
* Subject will receive a kidney with an anticipated cold ischemia time (CIT) of > 30 hours
* Recipient has a positive T or B-cell cross match by investigational site's standard method of determination
* Subject will receive a kidney from a 50-65 year old deceased donor with one of the following:

  * History of hypertension and a terminal serum creatinine > 1.5 mg/dL
  * Cerebrovascular accident as cause of death and a terminal serum creatinine > 1.5 mg/dL
  * History of hypertension and cerebrovascular accident as cause of death and a terminal serum creatinine > 1.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development; Principal Investigator, Principal Investigator — University of Michigan
Locations (38):
- United States (38):
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California - University Hospital, Los Angeles, California
  - St. Vincent/National Institute of Transplantation, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSD, San Diego, California
  - California Institute of Renal Research/Sharp Memorial Hospital, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Florida, Shands Hospital, Gainesville, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Medical College of Georgia, Augusta, Augusta, Georgia
  - Rush - Presbyterian - St. Lukes Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Buffalo General Hospital, Buffalo, New York
  - Mt. Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital - Cornell, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital of Cleveland, Cleveland, Ohio
  - Legacy Transplant Services, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Pinnacle Health at Harrisburg, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Methodist University Hospital - Memphis, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Methodist Hospital Research Institute of Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled de novo kidney transplant recipients who were at least 18 years of age.
Period: Overall Study
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Started | 82 | 80 | 80 | 81
Received Treatment | 79 | 77 | 75 | 78
Completed | 70 | 72 | 60 | 72
Not Completed | 12 | 8 | 20 | 9
Not completed — Death | 2 | 2 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Miscellaneous Reasons | 7 | 3 | 11 | 4
Not completed — Randomized but never received study drug | 3 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF | Total
Number analyzed (Participants) | 79 | 77 | 75 | 78 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.44 (15.077) | 49.26 (13.532) | 47.80 (12.469) | 49.68 (13.749) | 48.80 (13.707)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 27 | 24 | 99
  Male | 51 | 57 | 48 | 54 | 210

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biopsy-confirmed Acute Rejection (BCAR) at Month 6 Assessed by Local Review
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Biopsies were graded according to the 2005 Banff criteria. All biopsies (T-cell and/or antibody mediated) of grade 1 or higher were considered a BCAR.
  The Kaplan-Meier estimates at Day 182 was used for the analyses at 6 months. Lost to follow-up or patients with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants | 12.7 [6.5 to 18.9] | 26.3 [18.0 to 34.6] | 18.8 [11.4 to 26.3] | 16.7 [9.8 to 23.7]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Test type: Non-Inferiority or Equivalence — The aim of this study was to assess the non-inferiority of each experimental arm (Arms 2-4) to a comparator regimen (Arm 1) over a non-inferiority margin of 10%. If the upper bound of the 90% confidence interval was less than the margin, i.e., 10%, then the test treatment was considered to be non-inferior to the comparator regimen; Difference = 13.6, 90% CI 2-sided [3.2 to 23.9] — A positive difference indicates a higher failure rate in the experimental arm as compared to the comparator arm (Arm 1)
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 6.1, 90% CI 2-sided [-3.6 to 15.8] — A positive difference indicates a higher failure rate in the experimental arm as compared to the comparator arm (Arm 1)
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 4.0, 90% CI 2-sided [-5.3 to 13.3] — A positive difference indicated a higher failure rate in the experimental arm as compared to the comparator arm (Arm 1)

2. Secondary Outcome: Patient Survival at Month 6 and Month 12
Description: Patient survival is any participant who is known to be alive 6 months and 12 months after the skin closure date.
  The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 96.2 [92.7 to 99.7] | 94.8 [90.6 to 99.0] | 97.3 [94.3 to 100.0] | 93.6 [89.0 to 98.2]
  Month 12 | 87.3 [81.2 to 93.5] | 92.2 [87.2 to 97.2] | 87.8 [81.5 to 94.1] | 89.7 [84.1 to 95.4]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Patient survival at 6 months; Test type: Superiority or Other; Difference = -1.4, 90% CI 2-sided [-6.9 to 4.1]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Patient survival at 6 months; Test type: Superiority or Other; Difference = 1.1, 90% CI 2-sided [-3.5 to 5.8]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Patient survival at 6 months; Test type: Superiority or Other; Difference = -2.6, 90% CI 2-sided [-8.4 to 3.2]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Patient survival at 12 months; Test type: Superiority or Other; Difference = 4.9, 90% CI 2-sided [-3.1 to 12.8]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Patient survival at 12 months; Test type: Superiority or Other; Difference = 0.5, 90% CI 2-sided [-8.3 to 9.2]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Patient survival at 12 months; Test type: Superiority or Other; Difference = 2.4, 90% CI 2-sided [-6.0 to 10.8]

3. Secondary Outcome: Graft Survival at Month 6 and Month 12
Description: Graft survival was defined as any participant who was known to have a functioning graft (i.e., not graft loss) at 6 months and 12 months after the skin closure date. Graft loss was defined as patient death, retransplant, permanent return to dialysis (dialysis greater than 30 days) or transplant nephrectomy.
  The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 96.2 [92.7 to 99.7] | 93.5 [88.9 to 98.1] | 96.0 [92.3 to 99.7] | 92.3 [87.3 to 97.3]
  Month 12 | 87.3 [81.2 to 93.5] | 90.9 [85.5 to 96.3] | 86.5 [79.9 to 93.0] | 85.8 [79.2 to 92.3]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Graft survival at 6 months; Test type: Superiority or Other; Difference = -2.7, 90% CI 2-sided [-8.5 to 3.1]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Graft survival at 6 months; Test type: Superiority or Other; Difference = -0.2, 90% CI 2-sided [-5.3 to 4.9]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Graft survival at 6 months; Test type: Superiority or Other; Difference = -3.9, 90% CI 2-sided [-10.0 to 2.2]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Graft survival at 12 months; Test type: Superiority or Other; Difference = 3.6, 90% CI 2-sided [-4.6 to 11.7]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Graft survival at 12 months; Test type: Superiority or Other; Difference = -0.9, 90% CI 2-sided [-9.9 to 8.1]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Graft survival at 12 months; Test type: Superiority or Other; Difference = -1.6, 90% CI 2-sided [-10.6 to 7.4]

4. Secondary Outcome: Percentage of Participants With BCAR at Month 12 Assessed by Local Review
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Biopsies were graded according to the 2005 Banff criteria. All biopsies (T-cell and/or antibody mediated) of grade 1 or higher were considered a BCAR.
  The Kaplan-Meier estimates at Day 365 was used for the analyses at 12 months. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants | 15.4 [8.6 to 22.1] | 29.0 [20.4 to 37.6] | 20.2 [12.5 to 27.9] | 18.1 [10.9 to 25.3]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Test type: Superiority or Other; Difference = 13.7, 90% CI 2-sided [2.8 to 24.6]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Test type: Superiority or Other; Difference = 4.8, 90% CI 2-sided [-5.4 to 15.0]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Test type: Superiority or Other; Difference = 2.8, 90% CI 2-sided [-7.1 to 12.6]

5. Secondary Outcome: Percentage of Participants With BCAR at Month 6 and 12 Assessed by Central Review
Description: Rejection episodes were confirmed by biopsy by a central reviewer. Biopsies were graded according to the 2005 Banff criteria. All biopsies (T-cell and/or antibody mediated) of grade 1 or higher were considered a BCAR.
  The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 7.7 [2.7 to 12.7] | 18.3 [11.0 to 25.6] | 12.1 [5.9 to 18.3] | 14.2 [7.7 to 20.7]
  Month 12 | 7.7 [2.7 to 12.7] | 19.7 [12.2 to 27.2] | 12.1 [5.9 to 18.3] | 15.5 [8.8 to 22.3]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; BCAR at Month 6; Test type: Superiority or Other; Difference = 10.6, 90% CI 2-sided [1.8 to 19.5]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; BCAR at Month 6; Test type: Superiority or Other; Difference = 4.3, 90% CI 2-sided [-3.6 to 12.3]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; BCAR at Month 6; Test type: Superiority or Other; Difference = 6.4, 90% CI 2-sided [-1.7 to 14.6]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; BCAR at Month 12; Test type: Superiority or Other; Difference = 12.0, 90% CI 2-sided [3.0 to 21.0]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; BCAR at Month 12; Test type: Superiority or Other; Difference = 4.3, 90% CI 2-sided [-3.6 to 12.3]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; BCAR at Month 12; Test type: Superiority or Other; Difference = 7.8, 90% CI 2-sided [-0.6 to 16.2]

6. Secondary Outcome: Percentage of Participants With T-cell Mediated BCAR at Month 6 and 12 Assessed by Local Review
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Biopsies were graded according to the 2005 Banff criteria. All biopsies of grade 1 or higher were considered a BCAR.
  The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 12.7 [6.5 to 18.9] | 25.0 [16.8 to 33.1] | 18.8 [11.4 to 26.3] | 16.7 [9.8 to 23.7]
  Month 12 | 14.0 [7.6 to 20.5] | 27.7 [19.2 to 36.1] | 18.8 [11.4 to 26.3] | 18.1 [10.9 to 25.3]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 12.2, 90% CI 2-sided [2.0 to 22.5]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 6.1, 90% CI 2-sided [-3.6 to 15.8]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 4.0, 90% CI 2-sided [-5.3 to 13.3]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 13.6, 90% CI 2-sided [3.0 to 24.3]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 4.8, 90% CI 2-sided [-5.1 to 14.6]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 4.1, 90% CI 2-sided [-5.6 to 13.8]

7. Secondary Outcome: Percentage of Participants With T-cell Mediated BCAR at Month 6 and 12 Assessed by Central Review
Description: Rejection episodes were confirmed by biopsy by the central reviewer. Biopsies were graded according to the 2005 Banff criteria. All biopsies of grade 1 or higher were considered a BCAR.
  The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 7.7 [2.7 to 12.7] | 17.0 [9.9 to 24.1] | 12.1 [5.9 to 18.3] | 14.2 [7.7 to 20.7]
  Month 12 | 7.7 [2.7 to 12.7] | 18.4 [11.1 to 25.7] | 12.1 [5.9 to 18.3] | 15.5 [8.8 to 22.3]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 9.3, 90% CI 2-sided [0.7 to 18.0]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 4.3, 90% CI 2-sided [-3.6 to 12.3]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 6; Test type: Superiority or Other; Difference = 6.4, 90% CI 2-sided [-1.7 to 14.6]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 10.7, 90% CI 2-sided [1.8 to 19.5]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 4.3, 90% CI 2-sided [-3.6 to 12.3]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; T-cell Mediated BCAR at Month 12; Test type: Superiority or Other; Difference = 7.8, 90% CI 2-sided [-0.6 to 16.2]

8. Secondary Outcome: Change From Week 4 in Glomerular Filtration Rate Estimated by the MDRD Method at Month 6 and Month 12
Description: The glomerular filtration rate (GFR) was calculated using the Modification of Diet in Renal Disease (MDRD) method.
Time Frame: Week 4, Month 6 and Month 12
Population: Full analysis set with available data at Week 4. "N" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 71 | 66 | 70 | 72
mL/min per 1.73 m^2
  Week 4 | 54.7 (17.16) | 59.3 (24.01) | 51.6 (19.32) | 58.0 (16.97)
  Change at Month 6 (N=65, 66, 67, 66) | 5.7 (16.44) | 3.2 (13.86) | 8.3 (12.96) | 2.5 (12.82)
  Change at Month 12 (n=66, 64, 64, 66) | 8.9 (18.88) | 3.3 (16.55) | 9.1 (13.59) | 2.7 (16.60)

9. Secondary Outcome: Change From Week 4 in GFR by Iothalamate Clearance at Month 6
Description: The glomerular filtration rate was measured directly using iothalamate clearance.
Time Frame: Week 4 and Month 6
Population: Full analysis set with available data at Week 4. "N" indicates participants with available data at Week 4 and Month 6.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 59 | 49 | 50 | 55
mL/min per 1.73 m^2
  Week 4 | 48.00 (26.327) | 56.51 (33.612) | 44.36 (19.045) | 52.09 (25.696)
  Change at Month 6 (N=48, 45, 45, 47) | 5.81 (24.298) | 3.47 (34.708) | 3.56 (21.104) | 6.60 (35.090)

10. Secondary Outcome: Change From Week 4 in Serum Creatinine at Month 6 and 12
Time Frame: Week 4 and Month 6 and 12
Population: Full analysis set with available data at Week 4. "N" indicates participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 73 | 70 | 71 | 74
mg/dL
  Week 4 | 1.5 (0.68) | 1.6 (1.25) | 1.6 (0.84) | 1.5 (0.73)
  Change at Month 6 (N=69, 69, 68, 70) | -0.0 (0.64) | -0.2 (1.08) | -0.3 (0.64) | -0.0 (0.32)
  Change at Month 12 (N=67, 67, 65, 68) | -0.1 (0.45) | -0.2 (1.24) | -0.2 (0.76) | 0.1 (0.64)

11. Secondary Outcome: Percentage of Participants With Efficacy Failure at 6 and 12 Months Assessed by Local Review
Description: Efficacy failure is defined as death, graft failure (permanent return to dialysis [>30 days] or retransplant), BCAR according to local review, or lost to follow-up.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 15.2 [8.5 to 21.8] | 29.9 [21.3 to 38.4] | 22.7 [14.7 to 30.6] | 23.1 [15.2 to 30.9]
  Month 12 | 25.3 [17.3 to 33.4] | 33.8 [24.9 to 42.6] | 29.3 [20.7 to 38.0] | 29.5 [21.0 to 38.0]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 14.7, 90% CI 2-sided [3.8 to 25.5]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 7.5, 90% CI 2-sided [-2.9 to 17.8]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 7.9, 90% CI 2-sided [-2.4 to 18.2]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Efficacy Failure at Month12; Test type: Superiority or Other; Difference = 8.4, 90% CI 2-sided [-3.5 to 20.4]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Efficacy Failure at Month 12; Test type: Superiority or Other; Difference = 4.0, 90% CI 2-sided [-7.8 to 15.8]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Efficacy Failure at Month12; Test type: Superiority or Other; Difference = 4.2, 90% CI 2-sided [-7.5 to 15.9]

12. Secondary Outcome: Percentage of Participants With Efficacy Failure at 6 and 12 Months Assessed by Central Review
Description: Efficacy failure is defined as death, graft failure (permanent return to dialysis [>30 days] or retransplant), BCAR according to central review, or lost to follow-up.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 11.4 [5.5 to 17.3] | 22.1 [14.3 to 29.9] | 16.0 [9.0 to 23.0] | 20.5 [13.0 to 28.0]
  Month 12 | 19.0 [11.7 to 26.2] | 26.0 [17.8 to 34.2] | 21.3 [13.6 to 29.1] | 25.6 [17.5 to 33.8]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 10.7, 90% CI 2-sided [0.9 to 20.4]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 4.6, 90% CI 2-sided [-4.5 to 13.7]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Efficacy Failure at Month 6; Test type: Superiority or Other; Difference = 9.1, 90% CI 2-sided [-0.4 to 18.7]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Efficacy Failure at Month 12; Test type: Superiority or Other; Difference = 7.0, 90% CI 2-sided [-4.0 to 18.0]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Efficacy Failure at Month 12; Test type: Superiority or Other; Difference = 2.3, 90% CI 2-sided [-8.3 to 13.0]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Efficacy Failure at Month 12; Test type: Superiority or Other; Difference = 6.7, 90% CI 2-sided [-4.2 to 17.6]

13. Secondary Outcome: Time to First BCAR Assessed by Local Review
Description: The time to first BCAR (local review) was calculated as the first biopsy date in which the local reviewer confirmed an acute rejection minus the date of skin closure +1. Only participants with a BCAR are included in the analysis.
Time Frame: 12 months
Population: Full analysis set with a BCAR assessed by local review
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 12 | 22 | 15 | 14
days | 9 [5 to 194] | 12 [6 to 301] | 19 [7 to 195] | 12.5 [5 to 186]

14. Secondary Outcome: Time to First BCAR Assessed by Central Review
Description: The time to first BCAR (central review) was calculated as the first biopsy date in which the central reviewer confirmed an acute rejection minus the date of skin closure +1. Only participants with a BCAR are included in the analysis.
Time Frame: 12 months
Population: Full analysis set with a BCAR as assessed by the central reviewer
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 6 | 15 | 9 | 12
days | 19 [6 to 142] | 10 [7 to 187] | 12 [7 to 52] | 11.5 [5 to 295]

15. Secondary Outcome: Time to First T-cell Mediated BCAR Assessed by Local Review
Description: The time to first T-cell mediated BCAR (local review) was calculated as the first biopsy date in which the local reviewer confirmed an acute rejection minus the date of skin closure +1.
Time Frame: 12 months
Population: Full analysis set with a T-cell mediated BCAR as assessed by local review
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 11 | 21 | 14 | 14
days | 9 [5 to 194] | 12 [6 to 301] | 18 [7 to 178] | 12.5 [5 to 186]

16. Secondary Outcome: Time to First T-cell Mediated BCAR Assessed by Central Review
Description: The time to first T-cell mediated BCAR (central review) was calculated as the first biopsy date in which the central reviewer confirmed an acute rejection minus the date of skin closure +1. Only participants with a T-cell mediated BCAR are included in the analysis.
Time Frame: 12 months
Population: Full analysis set with a T-cell mediated BCAR as assessed by the central reviewer
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 6 | 14 | 9 | 12
days | 19 [6 to 142] | 10 [7 to 187] | 12 [7 to 52] | 11.5 [5 to 295]

17. Secondary Outcome: Maximum Grade of T-cell Mediated Rejection Assessed by Local Review
Description: The grade of acute T-cell mediated rejection was classified as IA, IB, IIA, IIB and III according to Banff 2005 criteria. If a patient had more than 1 T-cell mediated rejection, the episode with the most severe grade was used in the analysis.
  Grade IA: Cases with significant interstitial infiltration (> 25% of parenchyma affected) and foci of moderate tubulitis; Grade IB: Cases with significant interstitial infiltration (> 25% of parenchyma affected) and foci of severe tubulitis; Grade IIA: Cases with mild to moderate intimal arteritis; Grade IIB: Cases with severe intimal arteritis comprising >25% of the luminal area; Grade III: Cases with "transmural" arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
participants
  Month 6 - Grade IA | 4 | 6 | 8 | 2
  Month 6 - Grade IB | 3 | 4 | 3 | 4
  Month 6 - Grade IIA | 3 | 9 | 3 | 3
  Month 6 - Grade IIB | 0 | 0 | 0 | 4
  Month 6 - Grade III | 0 | 0 | 0 | 0
  Month 12 - Grade IA | 5 | 6 | 8 | 3
  Month 12 - Grade IB | 3 | 5 | 3 | 4
  Month 12 - Grade IIA | 3 | 10 | 3 | 3
  Month 12 - Grade IIB | 0 | 0 | 0 | 4
  Month 12 - Grade III | 0 | 0 | 0 | 0

18. Secondary Outcome: Maximum Grade of T-cell Mediated Rejection as Assessed by Central Review
Description: as for outcome 17
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
participants
  Month 6 - Grade IA | 1 | 1 | 2 | 1
  Month 6 - Grade IB | 0 | 3 | 1 | 1
  Month 6 - Grade IIA | 5 | 6 | 3 | 5
  Month 6 - Grade IIB | 0 | 2 | 3 | 4
  Month 6 - Grade III | 0 | 1 | 0 | 0
  Month 12 - Grade IA | 1 | 1 | 2 | 1
  Month 12 - Grade IB | 0 | 4 | 1 | 2
  Month 12 - Grade IIA | 5 | 6 | 3 | 5
  Month 12 - Grade IIB | 0 | 2 | 3 | 4
  Month 12 - Grade III | 0 | 1 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Clinically Treated Acute Rejection at Month 6 and Month 12
Description: Patients who received immunosuppressive medications for the treatment of suspected or BCAR were considered to have a clinically-treated acute rejection.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 19.0 [11.7 to 26.2] | 33.8 [24.9 to 42.6] | 29.3 [20.7 to 38.0] | 23.1 [15.2 to 30.9]
  Month 12 | 20.3 [12.8 to 27.7] | 35.1 [26.1 to 44.0] | 30.7 [21.9 to 39.4] | 23.1 [15.2 to 30.9]

20. Secondary Outcome: Percentage of Participants With Anti-lymphocyte-treated Rejection at Months 6 and 12
Description: Participants with histologically proved Banff Grade II or III rejection could receive anti-rejection therapy with anti-lymphocyte antibodies per institutional protocol.
  The use of anti-lymphocyte antibody therapy at any time during a suspected or proven rejection episode for the treatment of acute rejection was considered an event.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 6.3 [1.8 to 10.8] | 20.8 [13.2 to 28.4] | 12.0 [5.8 to 18.2] | 7.7 [2.7 to 12.7]
  Month 12 | 6.3 [1.8 to 10.8] | 20.8 [13.2 to 28.4] | 12.0 [5.8 to 18.2] | 7.7 [2.7 to 12.7]

21. Secondary Outcome: Percentage of Participants With Multiple Rejection Episodes at Months 6 and 12
Description: All participants were evaluated for the incidence of multiple rejection episodes (clinically treated and/or BCAR as assessed by the local reviewer) through 6 months and 12 months.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 1.3 [0.0 to 3.3] | 3.9 [0.3 to 7.5] | 4.0 [0.3 to 7.7] | 2.6 [0.0 to 5.5]
  Month 12 | 1.3 [0.0 to 3.3] | 7.8 [2.8 to 12.8] | 4.0 [0.3 to 7.7] | 3.8 [0.3 to 7.4]

22. Secondary Outcome: Percentage of Participants With Treatment Failure at Month 6 and 12
Description: Treatment failure was defined as death, graft loss, BCAR (local review), lost to follow-up or early discontinuation of treatment regimen. The Kaplan-Meier estimates at Days 182 and 365 were used for the analyses at 6 months and 12 months respectively. Lost to follow-up or participants with missing outcomes were censored at their last follow up visit.
Time Frame: 6 months and 12 months
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
percentage of participants
  Month 6 | 26.6 [18.4 to 34.8] | 37.7 [28.6 to 46.7] | 38.4 [29.0 to 47.7] | 29.5 [21.0 to 38.0]
  Month 12 | 35.5 [26.6 to 44.4] | 45.5 [36.1 to 54.8] | 45.2 [35.7 to 54.8] | 34.7 [25.8 to 43.6]
Statistical Analysis 1: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Treatment Failure at Month 6; Test type: Superiority or Other; Difference = 11.1, 90% CI 2-sided [-1.1 to 23.3]
Statistical Analysis 2: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Treatment Failure at Month 6; Test type: Superiority or Other; Difference = 11.8, 90% CI 2-sided [-0.7 to 24.2]
Statistical Analysis 3: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Treatment Failure at Month 6; Test type: Superiority or Other; Difference = 2.9, 90% CI 2-sided [-8.9 to 14.7]
Statistical Analysis 4: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus/MMF; Treatment Failure at Month 12; Test type: Superiority or Other; Difference = 10.0, 90% CI 2-sided [-2.9 to 22.8]
Statistical Analysis 5: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QW/Tacrolimus; Treatment Failure at Month 12; Test type: Superiority or Other; Difference = 9.7, 90% CI 2-sided [-3.3 to 22.8]
Statistical Analysis 6: Comparison: Tacrolimus/MMF/Basiliximab vs Alefacept QOW/Tacrolimus/MMF; Treatment Failure at Month 12; Test type: Superiority or Other; Difference = -0.8, 90% CI 2-sided [-13.3 to 11.7]

23. Secondary Outcome: Gastrointestinal Quality of Life Index Score Over Time
Description: The impact of gastrointestinal (GI) symptoms on health-related quality of life was assessed using the Gastrointestinal Quality of Life Index (GIQLI) symptom severity score. The GIQLI is a 36-item self-administered questionnaire that assesses the impact of gastrointestinal symptoms during the past 2 weeks on a scale from 0 (all of the time) to 4 (never). Possible overall scores ranged from 0 to 4, with higher scores indicating a better quality of life according to the different symptomatic criteria.
Time Frame: Months 1, 3, 6, and 12
Population: Full analysis set with available data at each time point (indicated by "N")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
units on a scale
  Month 1 (N=63, 60, 59, 58) | 2.85 (0.602) | 2.97 (0.541) | 3.00 (0.513) | 2.98 (0.493)
  Month 3 (N=53, 52, 53, 54) | 2.96 (0.595) | 3.29 (0.441) | 3.11 (0.516) | 3.16 (0.442)
  Month 6 (N=58, 61, 57, 59) | 3.05 (0.589) | 3.26 (0.450) | 3.24 (0.491) | 3.17 (0.456)
  Month 12 (N=62, 60, 52, 58) | 3.13 (0.524) | 3.18 (0.554) | 3.26 (0.605) | 3.19 (0.531)

24. Secondary Outcome: Gastrointestinal Symptom Rating Scale Scores Over Time
Description: The impact of gastrointestinal (GI) symptoms on health-related quality of life was assessed using the Gastrointestinal Symptom Rating Scale Scores (GSRS). The GSRS a 15-item self-administered questionnaire that assesses the impact of gastrointestinal symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort). Possible overall scores range from 1 to 7, with lower scores indicating a better quality of life with respect to gastrointestinal symptoms.
Time Frame: Months 1, 3, 6, and 12
Population: Full analysis set with available data at each time point (indicated by "N")
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Number analyzed (Participants) | 79 | 77 | 75 | 78
units on a scale
  Month 1 (N=70, 61, 61, 64) | 1.72 (0.665) | 1.43 (0.490) | 1.59 (0.674) | 1.48 (0.491)
  Month 3 (N=58, 55, 53, 56) | 1.52 (0.480) | 1.42 (0.672) | 1.47 (0.568) | 1.34 (0.370)
  Month 6 (N=63, 67, 62, 63) | 1.63 (0.602) | 1.41 (0.695) | 1.49 (0.471) | 1.42 (0.496)
  Month 12 (N=63, 65, 53, 65) | 1.63 (0.635) | 1.42 (0.564) | 1.52 (0.609) | 1.57 (0.642)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Tacrolimus/MMF/Basiliximab | Alefacept QW/Tacrolimus/MMF | Alefacept QW/Tacrolimus | Alefacept QOW/Tacrolimus/MMF
Serious Adverse Events (participants affected / at risk) | 41/79 | 48/77 | 40/75 | 45/78
Other Adverse Events (participants affected / at risk) | 79/79 | 77/77 | 75/75 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus/MMF/Basiliximab (N=79) | Alefacept QW/Tacrolimus/MMF (N=77) | Alefacept QW/Tacrolimus (N=75) | Alefacept QOW/Tacrolimus/MMF (N=78)
Urosepsis (Infections and infestations) | 3 | 2 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 3
Cytomegalovirus Viraemia (Infections and infestations) | 1 | 2 | 1 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 2 | 2 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 0
Polyomavirus-Associated Nephropathy (Infections and infestations) | 1 | 1 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 1 | 1 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 1 | 0 | 1
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 0 | 3 | 0
Aspergillosis (Infections and infestations) | 0 | 1 | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia Cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Arteriovenous Graft Site Infection (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
BK Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Catheter Related Infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis Enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis Of Male External Genital Organ (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridial Infection (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus Gastritis (Infections and infestations) | 0 | 1 | 0 | 0
Disseminated Cryptococcosis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Epstein-Barr Viraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia Infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter Gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1
Incision Site Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Intertrigo Candida (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis Cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Perinephric Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis Bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Herpes Viral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1 | 0
Retroperitoneal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis Syndrome (Infections and infestations) | 0 | 0 | 0 | 1
Skin Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Ureteritis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection Pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound Infection Bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 7 | 9 | 5 | 5
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 2
Renal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Perirenal Haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Post Procedural Urine Leak (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Graft Thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incision Site Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Renal Lymphocele (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transplant Failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Urinary Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Fluid Overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal Haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erosive Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0
Renal Vein Thrombosis (Renal and urinary disorders) | 1 | 1 | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 2 | 1 | 0
Focal Glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Nephritis Interstitial (Renal and urinary disorders) | 0 | 0 | 1 | 0
Obstructive Uropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Artery Thrombosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Mass (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Vasculitis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 4 | 4 | 2 | 5
Histology Abnormal (Investigations) | 0 | 1 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
Immunosuppressant Drug Level Increased (Investigations) | 1 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1
Urine Output Decreased (Investigations) | 0 | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 2 | 2
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Aortic Stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Renovascular Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Vascular Pseudoaneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 1 | 2
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 2 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 2
Angina Pectoris (Cardiac disorders) | 0 | 2 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 2 | 4
Chills (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anoxic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope Vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1
Unresponsive To Stimuli (Nervous system disorders) | 0 | 1 | 0 | 0
Removal Of Renal Transplant (Surgical and medical procedures) | 0 | 1 | 1 | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Pancreas Transplant (Surgical and medical procedures) | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Parathyroid Gland Enlargement (Endocrine disorders) | 0 | 1 | 0 | 0
Serum Sickness (Immune system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus/MMF/Basiliximab (N=79) | Alefacept QW/Tacrolimus/MMF (N=77) | Alefacept QW/Tacrolimus (N=75) | Alefacept QOW/Tacrolimus/MMF (N=78)
Anaemia (Blood and lymphatic system disorders) | 31 | 25 | 23 | 32
Leukocytosis (Blood and lymphatic system disorders) | 13 | 12 | 12 | 10
Leukopenia (Blood and lymphatic system disorders) | 13 | 23 | 13 | 16
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 5
Polycythaemia (Blood and lymphatic system disorders) | 4 | 3 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 1 | 5
Angina Pectoris (Cardiac disorders) | 6 | 2 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 3 | 5
Tachycardia (Cardiac disorders) | 8 | 13 | 10 | 9
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 3 | 11 | 10 | 11
Abdominal Pain (Gastrointestinal disorders) | 12 | 13 | 10 | 12
Abdominal Pain Lower (Gastrointestinal disorders) | 3 | 4 | 3 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2 | 3 | 6
Constipation (Gastrointestinal disorders) | 43 | 31 | 31 | 37
Diarrhoea (Gastrointestinal disorders) | 42 | 34 | 30 | 34
Dry Mouth (Gastrointestinal disorders) | 4 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 11 | 10 | 5 | 12
Dysphagia (Gastrointestinal disorders) | 3 | 4 | 3 | 2
Flatulence (Gastrointestinal disorders) | 2 | 5 | 4 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 10 | 6 | 5 | 7
Haemorrhoids (Gastrointestinal disorders) | 3 | 5 | 2 | 3
Nausea (Gastrointestinal disorders) | 52 | 37 | 39 | 42
Vomiting (Gastrointestinal disorders) | 24 | 18 | 15 | 16
Asthenia (General disorders) | 6 | 5 | 2 | 9
Catheter Site Pain (General disorders) | 2 | 4 | 1 | 0
Chills (General disorders) | 6 | 4 | 4 | 0
Fatigue (General disorders) | 12 | 16 | 18 | 12
Generalised Oedema (General disorders) | 3 | 3 | 5 | 3
Impaired Healing (General disorders) | 1 | 2 | 0 | 5
Oedema (General disorders) | 6 | 12 | 7 | 12
Oedema Peripheral (General disorders) | 27 | 22 | 28 | 31
Pain (General disorders) | 3 | 2 | 4 | 6
Pyrexia (General disorders) | 16 | 11 | 16 | 8
BK Virus Infection (Infections and infestations) | 15 | 16 | 17 | 20
Candiduria (Infections and infestations) | 0 | 0 | 4 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 3 | 4
Cytomegalovirus Viraemia (Infections and infestations) | 3 | 3 | 0 | 6
Escherichia Urinary Tract Infection (Infections and infestations) | 2 | 4 | 4 | 8
Nasopharyngitis (Infections and infestations) | 6 | 11 | 6 | 6
Oral Candidiasis (Infections and infestations) | 5 | 6 | 2 | 3
Sinusitis (Infections and infestations) | 2 | 8 | 5 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 16 | 10 | 9 | 8
Urinary Tract Infection (Infections and infestations) | 7 | 6 | 5 | 3
Urinary Tract Infection Bacterial (Infections and infestations) | 3 | 6 | 7 | 5
Urinary Tract Infection Enterococcal (Infections and infestations) | 2 | 3 | 4 | 6
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 11 | 18 | 9 | 19
Incision Site Complication (Injury, poisoning and procedural complications) | 2 | 4 | 4 | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 16 | 22 | 22 | 22
Perinephric Collection (Injury, poisoning and procedural complications) | 2 | 5 | 4 | 7
Post Procedural Discharge (Injury, poisoning and procedural complications) | 10 | 10 | 2 | 7
Procedural Nausea (Injury, poisoning and procedural complications) | 4 | 2 | 3 | 7
Procedural Pain (Injury, poisoning and procedural complications) | 63 | 58 | 51 | 64
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 4
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 15 | 4 | 10 | 2
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 4
Alanine Aminotransferase Increased (Investigations) | 1 | 4 | 1 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 6 | 3 | 2 | 3
Blood Creatinine Increased (Investigations) | 16 | 20 | 23 | 23
Blood Magnesium Decreased (Investigations) | 3 | 0 | 2 | 5
Blood Urea Increased (Investigations) | 1 | 4 | 2 | 2
CD4 Lymphocytes Decreased (Investigations) | 0 | 8 | 3 | 6
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 4 | 1 | 0
Immunosuppressant Drug Level Increased (Investigations) | 5 | 5 | 3 | 2
Liver Function Test Abnormal (Investigations) | 4 | 3 | 3 | 4
Transaminases Increased (Investigations) | 5 | 1 | 3 | 1
Urine Output Decreased (Investigations) | 2 | 5 | 3 | 3
Vitamin D Decreased (Investigations) | 2 | 5 | 2 | 0
Weight Increased (Investigations) | 9 | 7 | 9 | 11
White Blood Cell Count Increased (Investigations) | 4 | 1 | 3 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 6 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 5 | 5
Diabetes Mellitus (Metabolism and nutrition disorders) | 12 | 19 | 10 | 16
Fluid Overload (Metabolism and nutrition disorders) | 8 | 13 | 10 | 14
Fluid Retention (Metabolism and nutrition disorders) | 3 | 5 | 8 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 9 | 6 | 7 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 31 | 29 | 29
Hyperkalaemia (Metabolism and nutrition disorders) | 27 | 25 | 29 | 32
Hyperlipidaemia (Metabolism and nutrition disorders) | 11 | 7 | 8 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 7 | 6 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 14 | 20 | 14 | 25
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 7 | 5 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 27 | 15 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 | 32 | 38 | 44
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 8 | 6 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 32 | 39 | 36 | 38
Hypovolaemia (Metabolism and nutrition disorders) | 4 | 5 | 3 | 3
Metabolic Acidosis (Metabolism and nutrition disorders) | 11 | 12 | 4 | 7
Vitamin D Deficiency (Metabolism and nutrition disorders) | 15 | 7 | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 7 | 12 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 13 | 9
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 9 | 3 | 6
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 7 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 7 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 8 | 14 | 11
Dizziness (Nervous system disorders) | 12 | 11 | 12 | 11
Headache (Nervous system disorders) | 20 | 16 | 17 | 12
Hypoaesthesia (Nervous system disorders) | 2 | 5 | 4 | 2
Lethargy (Nervous system disorders) | 3 | 3 | 0 | 4
Paraesthesia (Nervous system disorders) | 3 | 4 | 5 | 1
Tremor (Nervous system disorders) | 34 | 18 | 35 | 20
Agitation (Psychiatric disorders) | 1 | 0 | 4 | 1
Anxiety (Psychiatric disorders) | 6 | 9 | 8 | 9
Depression (Psychiatric disorders) | 8 | 4 | 5 | 6
Insomnia (Psychiatric disorders) | 26 | 22 | 29 | 20
Bladder Spasm (Renal and urinary disorders) | 5 | 3 | 2 | 5
Dysuria (Renal and urinary disorders) | 9 | 6 | 12 | 8
Haematuria (Renal and urinary disorders) | 8 | 8 | 8 | 9
Hydronephrosis (Renal and urinary disorders) | 0 | 3 | 2 | 4
Nocturia (Renal and urinary disorders) | 2 | 4 | 0 | 2
Oliguria (Renal and urinary disorders) | 4 | 0 | 4 | 4
Pollakiuria (Renal and urinary disorders) | 4 | 4 | 3 | 1
Proteinuria (Renal and urinary disorders) | 7 | 6 | 10 | 8
Renal Tubular Necrosis (Renal and urinary disorders) | 2 | 7 | 5 | 3
Urinary Retention (Renal and urinary disorders) | 1 | 4 | 4 | 5
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 3 | 3 | 4
Erectile Dysfunction (Reproductive system and breast disorders) | 6 | 4 | 3 | 2
Scrotal Oedema (Reproductive system and breast disorders) | 3 | 4 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 14 | 10 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 14 | 14
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 3
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 14 | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 5
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7 | 1
Acne (Skin and subcutaneous tissue disorders) | 7 | 3 | 6 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7 | 4 | 8
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 15 | 15 | 14
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 6 | 5
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 4
Hypertension (Vascular disorders) | 35 | 32 | 29 | 31
Hypotension (Vascular disorders) | 12 | 15 | 12 | 15
Orthostatic Hypotension (Vascular disorders) | 7 | 1 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard Restriction Description: Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or 12 months after data-lock, whichever is first. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for up to 60 days to seek patent protection.